CLINICAL TRIAL: NCT03909126
Title: Pertussis Vaccination in Pregnant Women: Implementation and Evaluation of Different Models of Vaccination Dispensation
Brief Title: Pertussis Vaccination in Pregnant Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Collaborators: Ministere de la Sante et des Services Sociaux (Other)
Responsible Party: Principal Investigator, Caroline Quach, MD, Medical Lead Infection Prevention and Control, St. Justine's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MSSS-PERT-001
Record Dates: First submitted 2018-10-24; First posted 2019-04-09 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Pertussis
Keywords: pertussis; immunization coverage; vaccination; pregnant women; Quebec
MeSH Terms: conditions — Whooping Cough

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Montreal Region of Quebec (Experimental): Vaccination with Boostrix at time of gestational diabetes screening in a hospital setting
  Interventions: Biological: Boostrix administered during gestational diabetes screening
- Montérégie (No Intervention): Vaccination with Boostrix of pregnant women receiving routine care at the CLSC or regular clinic
- Maurice Region (Experimental): Vaccination with Boostrix of pregnant women receiving routine care at high volume clinic
  Interventions: Biological: Boostrix administered in high volume obstetric clinic
- National Capital (No Intervention): Vaccination with Boostrix of pregnant women receiving routine care at the CLSC or regular clinic

INTERVENTIONS:
Biological: Boostrix administered during gestational diabetes screening — Boostrix administered during gestational diabetes screening
  Arms: Montreal Region of Quebec
Biological: Boostrix administered in high volume obstetric clinic — Boostrix administered in high volume obstetric clinic
  Arms: Maurice Region

SUMMARY:
Brief Summary: The study compares four models of pertussis vaccination dispensation to pregnant women on the vaccine coverage obtained. In addition, the cost of the different models of vaccination will be evaluated.

DETAILED DESCRIPTION:
This is a quasi-experimental study with a non-equivalent control group in pregnant women, taking place in 4 regions of Québec (Montréal, Montérégie, Capitale-Nationale, Mauricie). Four models of vaccine dispensation will be evaluated: one university hospital around gestational diabetes screening, local health and social services centres (CSLC) and a high volume clinic. 250 participants will be recruited in each of the four types of centres.

In addition, the study will also evaluate the costs incurred by all those involved in the pertussis vaccination program for pregnant women as well as the cost per woman vaccinated.

Health Professionals:

15 to 20 health professionals involved in providing immunization services to pregnant women: obsterician-gynaecologists, family doctors and nurses in participating clinics will be interviewed to evaluate their knowledge, attitudes and professional practises regarding pertussis vaccination during pregnancy.

Evaluating the Cost:

A detailed costing approach (micro-costing) will be used. Time and movement will be studied by direct observation using a grid on an electronic file in each of the 5 environments studied in order to identify the services and activities carried out as well as to determine the resources involved in the implementation of these services and activities. Three typical vaccination days will be chosen to make these observations, in each of the four study environments.

The main activities observed will be related to preparations for vaccination up to the vaccination itself (informed consent, injection, etc.), the capture of vaccination data the management of vaccines and equipment, clinical manifestations, etc. If necessary, the people observed can be interviewed directly to better understand the activities or services provided. Otherwise, some questions may be included in the interviews described above.

The major cost categories that will be evaluated for each of the delivery modalities are human resources and supplies. The cost components listed are: nursing time (immunization / training), coordination time, support staff time, office supplies, vaccine storage equipment, vaccine transportation equipment, vaccine transportation, health and safety equipment, emergency, single-use vaccination equipment and others.

With regard to the costs borne by women, the main categories of variables evaluated will be: the time spent making appointments and attending vaccination appointments, working time lost, if any, transportation, childcare and other expenses

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women at least 18 years old who speak English or French
* Signed Informed Consent

Exclusion Criteria:

-

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant females
Enrollment: 946 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
Proportion of pregnant women vaccinated against pertussis | 11 months, May 2019 o March 2020
  Proportion of pregnant women vaccinated against pertussis will be evaluated in 5 Quebec regions
Proportion of pregnant women who consider pertussis as serious risk for infant | 12 months, May 2019 to April 2020
  Understanding of pertussis risk
Proportion of pregnant women who consider pertussis vaccination during pregnancy as safe. | 12 months, May 2019 to April 2020
  Understanding of vaccine risk perception in pregnant women
Costs for each vaccinated woman | 12 months, January to December 2019
  The cost of vaccination will be evaluated and compared between the four vaccination models.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Quach, MD, Principal Investigator — St. Justine's Hospital
Locations (3):
- Canada (3):
  - CLSC Montérégie, Longueuil, Quebec
  - CHU Sainte-Justine, Montreal, Quebec
  - CLSC Capitale Nationale, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No